CLINICAL TRIAL: NCT02918968
Title: A Randomized Phase IV Study Comparing Enzalutamide Versus Flutamide in Castration-resistant Prostate Cancer (CRPC) Patients Who Have Failed Combined Androgen Blockade Therapy With Bicalutamide Plus Androgen Deprivation Therapy (ADT)
Brief Title: Study on Enzalutamide and Flutamide in Patients With Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9785-MA-3051
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Results first posted 2021-05-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: enzalutamide; Xtandi; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Flutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enzalutamide 160 mg 1st line AAT/Flutamide 375 mg 2nd line AAT (Experimental): Participants received enzalutamide 160 mg capsules, orally once daily as 1st line of alternative antiandrogen therapy (AAT) until confirmed prostate-specific antigen (PSA) progression, other disease progression, or an intolerable adverse event. After confirmation of PSA progression, other disease progression, or an intolerable adverse event, participants received flutamide 125 mg tablets orally thrice daily after each meal as 2nd line of AAT. Treatment with each drug was continued until the participant met any of the discontinuation criteria or until 2 years from the enrollment of the last participant (approximately 38 months).
  Interventions: Drug: Enzalutamide; Drug: Flutamide; Other: Androgen deprivation therapy
- Flutamide 375 mg 1st line AAT/Enzaltumide 160 mg 2nd line AAT (Experimental): Participants received flutamide 125 mg tablets orally thrice daily after each meal as 1st line of AAT until confirmed PSA progression, other disease progression, or an intolerable adverse event. After confirmed PSA progression, other disease progression, or an intolerable adverse event. participants received enzalutamide 160 mg capsules orally once daily as 2nd line of AAT. Treatment with each drug was continued until the participant met any of the discontinuation criteria or until 2 years from the enrollment of the last participant (approximately 38 months).
  Interventions: Drug: Enzalutamide; Drug: Flutamide; Other: Androgen deprivation therapy

INTERVENTIONS:
Drug: Enzalutamide — Oral Capsule
  Other Names: Xtandi; MDV3100
Drug: Flutamide — Oral tablet
Other: Androgen deprivation therapy — All subjects must undergo continuous Androgen deprivation therapy with GnRH agonist/antagonist or bilateral orchiectomy during the study period.

SUMMARY:
The objective of this study was to compare the efficacy and safety of the combination therapy with enzalutamide + androgen deprivation therapy (ADT) and the combination therapy with flutamide + ADT in patients with castration resistant prostate cancer who had relapsed during combined androgen blockade (CAB) therapy with bicalutamide and ADT. This study also investigated the order of alternative antiandrogen therapy (AAT) by changing the 1st line medication after relapse of prostate-specific antigen (PSA).

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small-cell histology.
* Subject on continuous ADT with Gonadotropin Releasing Hormone (GnRH) agonist/antagonist or bilateral orchiectomy.
* Serum testosterone level below the target level at screening visit.
* Subject with asymptomatic or mildly symptomatic prostate cancer.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject has progression of the disease as defined by rising PSA levels or progressive soft tissue or bony disease during CAB therapy in combination of bicalutamide and ADT.
* A sexually active male subject and the subject's female partner who is of childbearing potential must use 2 acceptable birth control methods from screening to 3 months after the last dose of the study drug.
* Subject must agree not to donate sperm from screening to 3 months after the last dose of the study drug.

Exclusion Criteria:

* Subject with severe concurrent diseases, infections, or complications.
* Subject with confirmed or suspected brain metastasis or active leptomeningeal metastasis.
* Subject with a history of malignant tumor other than prostate cancer in the past 5 years.
* Subject hypersensitive to the ingredients of enzalutamide capsules or flutamide tablets.
* Subject with a history of convulsive attack, or prone to convulsive attack.
* Subject with liver disorder such as viral hepatitis and hepatic cirrhosis, or subject with Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) at screening visit higher than the upper limit of normal.
* Subject received treatment for prostate cancer with cytocidal chemotherapy that includes anti androgenic agents other than bicalutamide, abiraterone, or estramustine.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (47):
- Japan (47):
  - Site JP00024, Nagoya, Aichi-ken
  - Site JP00025, Nagoya, Aichi-ken
  - Site JP00038, Matsuyama, Ehime
  - Site JP00051, Iizuka, Fukuoka
  - Site JP00045, Isesaki, Gunma
  - Site JP00005, Maebashi, Gunma
  - Site JP00043, Ōta, Gunma
  - Site JP00054, Hakodate, Hokkaido
  - Site JP00001, Sapporo, Hokkaido
  - Site JP00002, Sapporo, Hokkaido
  - Site JP00048, Sapporo, Hokkaido
  - Site JP00055, Mito, Ibaraki
  - Site JP00019, Sagamihara, Kanagawa
  - Site JP00020, Yokohama, Kanagawa
  - Site JP00021, Yokohama, Kanagawa
  - Site JP00044, Yokosuka, Kanagawa
  - Site JP00046, Kashihara, Nara
  - Site JP00033, Kurashiki, Okayama-ken
  - Site JP00028, Hirakata, Osaka
  - Site JP00030, Sayama, Osaka
  - Site JP00027, Suita, Osaka
  - Site JP00009, Kitaadachi-gun, Saitama
  - Site JP00022, Hamamatsu, Shizuoka
  - Site JP00049, Utsunomiya, Tochigi
  - Site JP00011, Bunkyo-ku, Tokyo
  - Site JP00017, Bunkyo-ku, Tokyo
  - Site JP00013, Koto-ku, Tokyo
  - Site JP00014, Nakano-ku, Tokyo
  - Site JP00016, Shinagawa-ku, Tokyo
  - Site JP00018, Shinjuku-ku, Tokyo
  - Site JP00034, Ube, Yamaguchi
  - Site JP00010, Chiba
  - Site JP00053, Chiba
  - Site JP00039, Fukuoka
  - Site JP00040, Fukuoka
  - Site JP00050, Fukuoka
  - Site JP00035, Hiroshima
  - Site JP00026, Kyoto
  - Site JP00006, Nagano
  - Site JP00008, Nagano
  - Site JP00041, Nagasaki
  - Site JP00029, Osaka
  - Site JP00031, Osaka
  - Site JP00032, Osaka
  - Site JP00042, Saga
  - Site JP00037, Tokushima
  - Site JP00052, Toyama

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=402
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217491&parentIdentifier=9785-MA-3051&attachmentIdentifier=f355cf0d-cc7a-43df-bbfa-a7e32208d80a&fileName=9785-MA-3051_Plain_language_summary_JP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with M0 or M1 castration-resistant prostatic neoplasm that relapsed during Combined Androgen Blockade (CAB) therapy with bicalutamide were enrolled in this study.
Pre-assignment Details: Randomization was stratified by disease stages (M0/N0, M0/N1 or M1).
Groups:
- Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT: Participants received enzalutamide 160 mg capsules, orally once daily as 1st line of alternative antiandrogen therapy (AAT) until confirmed prostate-specific antigen (PSA) progression, other disease progression, or an intolerable adverse event. After confirmed PSA progression, other disease progression, or an intolerable adverse event, participants received flutamide 125 mg tablets orally thrice daily after each meal as 2nd line of AAT. Treatment with each drug was continued until the participant met any of the discontinuation criteria or until 2 years from the enrollment of the last participant (approximately 38 months).
- Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT: Participants received flutamide 125 mg tablets orally thrice daily after each meal as 1st line of AAT until confirmed PSA progression, other disease progression, or an intolerable adverse event. After confirmed PSA progression, other disease progression, or an intolerable adverse event, participants received enzalutamide 160 mg capsules orally once daily as 2nd line of AAT. Treatment with each drug was continued until the participant met any of the discontinuation criteria or until 2 years from the enrollment of the last participant (approximately 38 months).
Period: 1st Line AAT
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Started | 102 | 104
Maintained 1st Line AAT Without Progression | 25 | 8
Completed | 73 | 93
Not Completed | 29 | 11
Not completed — Progressive disease | 9 | 4
Not completed — Adverse Event | 12 | 3
Not completed — Physician Decision | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 0
Not completed — Miscellaneous | 1 | 0
Period: 2nd Line AAT
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Started | 48 (Participants who maintained 1st line AAT without progression did not enter 2nd line AAT) | 85 (Participants who maintained 1st line AAT without progression did not enter 2nd line AAT)
Completed | 23 | 73
Not Completed | 25 | 12
Not completed — Progressive disease | 21 | 3
Not completed — Adverse Event | 2 | 5
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population was defined as all participants randomized in this study.
Groups:
- Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT: Participants received enzalutamide 160 mg capsules, orally once daily as 1st line of AAT until confirmed PSA progression, other disease progression, or an intolerable adverse event. After confirmed PSA progression, other disease progression, or an intolerable adverse event, participants received flutamide 125 mg tablets orally thrice daily after each meal as 2nd line of AAT. Treatment with each drug was continued until the participant met any of the discontinuation criteria or until 2 years from the enrollment of the last participant (approximately 38 months).
- Total: Total of all reporting groups
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (7.6) | 74.1 (7.6) | 74.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 102 | 104 | 206
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease Stages at Randomization [Number; unit: Participants] — Number of participants in each disease stage (M0/N0, M0/N1, M1) at randomization were reported. 1) M0/N0: No distant metastasis and no lymph node metastasis. 2) M0/N1: Without distant metastasis, but with metastasis in lymph nodes distal to the aortic bifurcation. 3) M1: With distant metastasis (including metastasis in lymph nodes proximal to the aortic bifurcation).
  Participants
    M0/N0 | 24 | 25 | 49
    M0/N1 | 3 | 4 | 7
    M1 | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Time to PSA Progression With 1st Line AAT (TTPP1)
Description: TTPP1 was defined as the period from the date of randomization to the date of PSA progression in the 1st line AAT period. PSA progression was defined according to the consensus guidelines of prostate cancer clinical trials working group 2 (PCWG2). For participants with PSA declines at week 13, the PSA progression date was defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir were documented, which was confirmed by a second consecutive value obtained 3 or more weeks later. For participants with no PSA decline at week 13, the PSA progression date was defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the baseline were documented. Time to event analysis was performed using kaplan-meier (KM) estimates.
Time Frame: From date of randomization to the date of PSA progression in the 1st line AAT period (Up to 38 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 102 | 104
Months | 21.39 [12.16 to NA] — Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5. | 5.78 [4.67 to 8.54]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; Test type: Superiority — The significance level was 0.05 (two-sided); p < 0.001, Log Rank — P-value is based on a log-rank test stratified disease stages (M0/N0, M0/N1, or M1); Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.29 to 0.61] — Hazard ratio and P-value calculated using unstratified Cox proportional hazards model with treatment and disease stages (M0/N0, M0/N1, or M1) as covariate

2. Secondary Outcome: Time to PSA Progression With 2nd Line AAT (TTPP2)
Description: TTPP2 was defined as the period from day 1 of the 2nd line AAT to the date of PSA progression with the 2nd line AAT. PSA progression was defined according to the consensus guidelines of PCWG2. For participants with PSA declines at week 13, the PSA progression date was defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir were documented, which was confirmed by a second consecutive value obtained 3 or more weeks later. For participants with no PSA decline at week 13, the PSA progression date was defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the baseline were documented. Time to event analysis was performed using kaplan-meier estimates.
Time Frame: From date of randomization to the date of PSA progression in 2nd line AAT (Up to 38 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 102 | 104
Months | NA [20.99 to NA] — Median was not estimable since KM estimate did not reach to 50%. Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5. | 21.22 [14.78 to NA] — Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5.

3. Secondary Outcome: Percentage of Participants Achieving at Least 50 or 90 Percent (%) Reduction From Baseline and Up To Week 38 in Prostate Specific Antigen (PSA) Response at 1st Line AAT
Description: PSA response was defined as PSA decreased by at least 50% or 90% from baseline when at least 3 weeks passed after the lowest PSA decreased by at least 50% or 90% from baseline in the 1st line AAT period after baseline.
  Data was reported per each disease stage (M0/N0, M0/N1, M1). 1) M0/N0: No distant metastasis and no lymph node metastasis. 2) M0/N1: Without distant metastasis, but with metastasis in lymph nodes distal to the aortic bifurcation. 3) M1: With distant metastasis (including metastasis in lymph nodes proximal to the aortic bifurcation).
Time Frame: Baseline and at least 3 weeks after, the lowest PSA decreased by at least 50% or 90% from baseline (Up to 38 months)
Population: ITT population with participants in each disease stage.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 102 | 104
Percentage of participants
  M0/N0: (≥ 50% reduction): number analyzed (Participants) | 24 | 25
  M0/N0: (≥ 50% reduction) | 75.0 [53.3 to 90.2] | 48.0 [27.8 to 68.7]
  M0/N1: (≥ 50% reduction): number analyzed (Participants) | 3 | 4
  M0/N1: (≥ 50% reduction) | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 60.2]
  M1: (≥ 50% reduction): number analyzed (Participants) | 75 | 75
  M1: (≥ 50% reduction) | 72.0 [60.4 to 81.8] | 32.0 [21.7 to 43.8]
  All participants: (≥ 50% reduction) | 72.5 [62.8 to 80.9] | 34.6 [25.6 to 44.6]
  M0/N0: (≥ 90% reduction): number analyzed (Participants) | 24 | 25
  M0/N0: (≥ 90% reduction) | 62.5 [40.6 to 81.2] | 8.0 [1.0 to 26.0]
  M0/N1: (≥ 90% reduction): number analyzed (Participants) | 3 | 4
  M0/N1: (≥ 90% reduction) | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 60.2]
  M1: (≥ 90% reduction): number analyzed (Participants) | 75 | 75
  M1: (≥ 90% reduction) | 53.3 [41.4 to 64.9] | 20.0 [11.6 to 30.8]
  All participants: (≥ 90% reduction) | 54.9 [44.7 to 64.8] | 16.3 [9.8 to 24.9]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; >=50% reduction; Test type: Superiority — The significance level was 0.05 (two-sided); p < 0.001, Mantel Haenszel — P-value is based on Cochran-Mantel-Haenszel mean score test stratified disease stages (M0/N0, M0/N1, or M1); Mantel Haenszel common risk difference; Risk Difference (RD) = 37.8, 95% CI 2-sided [25.2 to 50.4] — Difference of response rate
Statistical Analysis 2: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; ≥ 90% reduction; Test type: Superiority — The significance level was 0.05 (two-sided); p < 0.001, Mantel Haenszel — P-value is based on Cochran-Mantel-Haenszel mean score test stratified disease stages (M0/N0, M0/N1, or M1); Mantel Haenszel common risk difference; Risk Difference (RD) = 38.4, 95% CI 2-sided [26.3 to 50.4] — Difference of response rate

4. Secondary Outcome: Percentage of Participants Achieving at Least 50 or 90 Percent (%) Reduction From Baseline to Week 13 in Prostate Specific Antigen (PSA) Response at 1st Line AAT
Description: PSA response was defined as the lowest PSA at week 13 decreased by at least 50% or 90% from baseline in the 1st line AAT period.
  Data was reported per each disease stage (M0/N0, M0/N1, M1). 1) M0/N0: No distant metastasis and no lymph node metastasis. 2) M0/N1: Without distant metastasis, but with metastasis in lymph nodes distal to the aortic bifurcation. 3) M1: With distant metastasis (including metastasis in lymph nodes proximal to the aortic bifurcation).
Time Frame: Baseline and week 13
Population: ITT population with participants in each disease stage.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 102 | 104
Percentage of participants
  M0/N0: (≥ 50% reduction): number analyzed (Participants) | 24 | 25
  M0/N0: (≥ 50% reduction) | 83.3 [62.6 to 95.3] | 40.0 [21.1 to 61.3]
  M0/N1: (≥ 50% reduction): number analyzed (Participants) | 3 | 4
  M0/N1: (≥ 50% reduction) | 66.7 [9.4 to 99.2] | 0.0 [0.0 to 60.2]
  M1: (≥ 50% reduction): number analyzed (Participants) | 75 | 75
  M1: (≥ 50% reduction) | 72.0 [60.4 to 81.8] | 33.3 [22.9 to 45.2]
  All participants: (≥ 50% reduction) | 74.5 [64.9 to 82.6] | 33.7 [24.7 to 43.6]
  M0/N0: (≥ 90% reduction): number analyzed (Participants) | 24 | 25
  M0/N0: (≥ 90% reduction) | 50.0 [29.1 to 70.9] | 8.0 [1.0 to 26.0]
  M0/N1: (≥ 90% reduction): number analyzed (Participants) | 3 | 4
  M0/N1: (≥ 90% reduction) | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 60.2]
  M1: (≥ 90% reduction): number analyzed (Participants) | 75 | 75
  M1: (≥ 90% reduction) | 49.3 [37.6 to 61.1] | 18.7 [10.6 to 29.3]
  All participants: (≥ 90% reduction) | 49.0 [39.0 to 59.1] | 15.4 [9.1 to 23.8]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; ≥ 50% reduction; Test type: Superiority — The significance level was 0.05 (two-sided); p < 0.001, Mantel Haenszel — P-value is based on Cochran-Mantel-Haenszel mean score test stratified disease stages (M0/N0, M0/N1, or M1); Mantel Haenszel common risk difference; Risk Difference (RD) = 40.7, 95% CI 2-sided [28.3 to 53.1] — Difference of response rate
Statistical Analysis 2: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; ≥90% reduction; Test type: Superiority — The significance level was 0.05 (two-sided); p < 0.001, Mantel Haenszel — P-value is based on Cochran-Mantel-Haenszel mean score test stratified disease stages (M0/N0, M0/N1, or M1); Mantel Haenszel common risk difference; Risk Difference (RD) = 33.5, 95% CI 2-sided [21.5 to 45.4] — Difference of response rate

5. Secondary Outcome: Time to PSA Decrease by 50% From Baseline With 1st Line AAT
Description: Time to PSA decrease by 50% with 1st line AAT was defined as the period from the date of randomization to the day when the decrease of PSA from baseline by 50% is first identified. Time to event analysis was performed using kaplan-meier estimates.
  Data was reported per each disease stage (M0/N0, M0/N1, M1). 1) M0/N0: No distant metastasis and no lymph node metastasis. 2) M0/N1: Without distant metastasis, but with metastasis in lymph nodes distal to the aortic bifurcation. 3) M1: With distant metastasis (including metastasis in lymph nodes proximal to the aortic bifurcation).
Time Frame: From date of randomization to the day when the decrease of PSA from baseline by 50% is first identified (Up to 38 months)
Population: ITT population with participants in each disease stage.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 102 | 104
Months
  M0/N0: number analyzed (Participants) | 24 | 25
  M0/N0 | 2.79 [2.66 to 3.02] | 3.94 [2.79 to NA] — Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5.
  M0/N1: number analyzed (Participants) | 3 | 4
  M0/N1 | 2.79 [2.56 to NA] — Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5. | NA [NA to NA] — Median was not estimable since KM estimate did not reach to 50%. Lower limit of confidence interval was not estimable since the lower confidence limits for the survivor function lay above 0.5. Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5.
  M1: number analyzed (Participants) | 75 | 75
  M1 | 2.79 [NA to NA] — Lower and upper limit of confidence interval were not estimable since a lot of participants had event at same study day. | 7.49 [3.02 to NA] — Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5.
Statistical Analysis 1: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; Test type: Superiority — The significance level was 0.05 (two-sided); p < 0.001, Log Rank — P-value is based on a log-rank test stratified disease stages (M0/N0, M0/N1, or M1)

6. Secondary Outcome: Time to Treatment Failure of 1st Line AAT (TTF1)
Description: TTF1 was defined as the period from randomization to study drug discontinuation of 1st line AAT for any reason that includes disease progression, onset of adverse events (AEs), participants request, or death. Time to event analysis was performed using kaplan-meier estimates.
  Data was reported per each disease stage (M0/N0, M0/N1, M1). 1) M0/N0: No distant metastasis and no lymph node metastasis. 2) M0/N1: Without distant metastasis, but with metastasis in lymph nodes distal to the aortic bifurcation. 3) M1: With distant metastasis (including metastasis in lymph nodes proximal to the aortic bifurcation).
Time Frame: From date of randomization to discontinuation of 1st line AAT (Up to 38 months)
Population: ITT population with participants in each disease stage.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 102 | 104
Months
  M0/N0: number analyzed (Participants) | 24 | 25
  M0/N0 | 17.58 [10.15 to 24.11] | 7.72 [4.47 to 15.67]
  M0/N1: number analyzed (Participants) | 3 | 4
  M0/N1 | 5.55 [4.86 to 10.38] | 4.73 [1.87 to 7.62]
  M1: number analyzed (Participants) | 75 | 75
  M1 | 12.02 [7.39 to 18.43] | 3.94 [3.65 to 5.55]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; Test type: Superiority — The significance level was 0.05 (two-sided); p < 0.001, Log Rank — P-value is based on a log-rank test stratified disease stages (M0/N0, M0/N1, or M1)

7. Secondary Outcome: Time to Treatment Failure of 2nd Line AAT (TTF2)
Description: TTF2 was defined as the period from randomization to study drug discontinuation of 2nd line AAT for any reason that includes disease progression, onset of AEs, participants request, or death. Time to event analysis was performed using kaplan-meier estimates.
Time Frame: From date of randomization to discontinuation of 2nd line AAT (Up to 38 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 102 | 104
Months | 23.03 [16.79 to NA] — Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5. | 16.59 [13.14 to 23.95]

8. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Description: rPFS was defined as the period from randomization to the time when radiographic disease progression is observed or death of any cause during the study period, whichever occurs earlier. Time to event analysis was performed using kaplan-meier estimates.
  Data was reported per each disease stage (M0/N0, M0/N1, M1). 1) M0/N0: No distant metastasis and no lymph node metastasis. 2) M0/N1: Without distant metastasis, but with metastasis in lymph nodes distal to the aortic bifurcation. 3) M1: With distant metastasis (including metastasis in lymph nodes proximal to the aortic bifurcation).
Time Frame: From date of randomization to the time when radiographic disease progression is observed or death of any cause (up to 38 months)
Population: ITT population with M1 diseases stage participants. No data reported for M0/N0 and M0/N1 as there are zero participants with event.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT | Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT
Number analyzed (Participants) | 75 | 104
Months
  M0/N0: number analyzed (Participants) | 0 | 0
  M0/N1: number analyzed (Participants) | 0 | 0
  M1 | NA [NA to NA] — Median was not estimable since KM estimate did not reach to 50%. Lower limit of confidence interval was not estimable since the lower confidence limits for the survivor function lay above 0.5. Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5. | NA [29.08 to NA] — Median was not estimable since KM estimate did not reach to 50%. Upper limit of confidence interval was not estimable since the upper confidence limits for the survivor function lay above 0.5.
Statistical Analysis 1: Comparison: Enzalutamide 160 mg 1st Line AAT/Flutamide 375 mg 2nd Line AAT vs Flutamide 375 mg 1st Line AAT/Enzaltumide 160 mg 2nd Line AAT; Test type: Superiority — The significance level was 0.05 (two-sided); p = 0.669, Log Rank — P-value is based on a log-rank test stratified disease stages (M0/N0, M0/N1, or M1); Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.45 to 1.67] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From of date of randomization to end of study (up to 38 months)
Groups:
- Enzalutamide 160mg 1st Line AAT: Participants received enzalutamide 160mg capsules orally once daily as 1st line of AAT until confirmed PSA progression, other disease progression, or an intolerable adverse event (approximately 38 months).
- Enzalutamide 160mg 2nd Line AAT: Participants received enzalutamide 160mg capsules orally once daily as 2nd line of AAT after confirmed PSA progression, other disease progression, or an intolerable adverse event (approximately 38 months).
- Flutamide 375mg 1st Line AAT: Participants received flutamide 125mg tablets orally thrice daily after each meal as 1st line of AAT until confirmed PSA progression, other disease progression, or an intolerable adverse event (approximately 38 months).
- Flutamide 375mg 2nd Line AAT: Participants received flutamide 125mg tablets orally thrice daily as 2nd line of AAT after confirmed PSA progression, other disease progression, or an intolerable adverse event (approximately 38 months).
Arm/Group | Enzalutamide 160mg 1st Line AAT | Enzalutamide 160mg 2nd Line AAT | Flutamide 375mg 1st Line AAT | Flutamide 375mg 2nd Line AAT
All-Cause Mortality (participants affected / at risk) | 1/102 | 1/85 | 0/104 | 0/48
Serious Adverse Events (participants affected / at risk) | 29/102 | 18/85 | 15/104 | 4/48
Other Adverse Events (participants affected / at risk) | 79/102 | 56/85 | 65/104 | 22/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide 160mg 1st Line AAT (N=102) | Enzalutamide 160mg 2nd Line AAT (N=85) | Flutamide 375mg 1st Line AAT (N=104) | Flutamide 375mg 2nd Line AAT (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Malignant neoplasm papilla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mental fatigue (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric calculus removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide 160mg 1st Line AAT (N=102) | Enzalutamide 160mg 2nd Line AAT (N=85) | Flutamide 375mg 1st Line AAT (N=104) | Flutamide 375mg 2nd Line AAT (N=48)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 14 (16) | 2 (2) | 3 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 5 (5) | 7 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (3) | 12 (14) | 6 (6)
Nausea (Gastrointestinal disorders) | 7 (8) | 6 (7) | 5 (5) | 2 (2)
Fatigue (General disorders) | 15 (17) | 8 (10) | 3 (3) | 0 (0)
Malaise (General disorders) | 15 (16) | 17 (19) | 4 (4) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 2 (2) | 9 (10) | 2 (2)
Influenza (Infections and infestations) | 7 (7) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 23 (36) | 12 (17) | 17 (33) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 18 (21) | 10 (10) | 4 (4) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 7 (8) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 6 (7) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 8 (9) | 4 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 4 (4) | 6 (6) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 6 (6) | 5 (5) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 6 (6) | 2 (2) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 4 (4) | 1 (1) | 6 (6) | 0 (0)
Hypertension (Vascular disorders) | 13 (15) | 5 (6) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT02918968/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02918968/SAP_001.pdf